CLINICAL TRIAL: NCT05562102
Title: An Open-label Effectiveness Study of a Typhoid Conjugate Vaccine in Kisantu, Democratic Republic of Congo (TyVECO) - Step 3: Surveillance Protocol
Brief Title: TyVECO: Surveillance Protocol
Acronym: TyVECO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Vaccine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-004
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-08

CONDITIONS: Typhoid Fever; Intestinal Perforation
MeSH Terms: conditions — Typhoid Fever; Intestinal Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Typbar-TCV, Bharat Biotech — Typhoid conjugate vaccine

SUMMARY:
In Kisantu Health Zone, approximate population 200,000, fever surveillance will be implemented in 8 health centers and 1 tertiary hospital. Individuals presenting to one of these study facilities with acute fever or history of fever or individuals presenting with suspicion of intestinal perforation irrespective of fever status, will be considered for enrollment. Following consent, blood samples (between 2.5 ml for children and 22 ml for adults) will be collected from eligible subjects and demographic and clinical information will be recorded in study forms at the time of enrollment at study health centers and hospitals. Peritoneal fluid and ileal tissue samples will be collected from surgical patients where possible. Biological specimens will be used for various testing, including microbiological culture of blood, tissue and peritoneal fluid for confirmation of bacterial growth, malaria diagnostics (microscopy and rapid testing), and storage of tissue samples for pathological investigation, and biobanking. Hospitalized patients will be followed-up to track clinical outcomes for the duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

At health center:

1. Patients of all ages currently living in the catchment area of the health center presenting to healthcare facility with objective fever of at least 38.0°C tympanic or 37.5 °C axillary OR
2. Patients of all ages currently living in the catchment area of the health center presenting to healthcare facility with reported fever ≥3 consecutive days within 7 days of presentation

At Hospital:

1. Suspicion of intestinal perforation/peritonitis due to typhoid fever requiring surgery for patients living in and outside the catchment area (even in the absence of laboratory confirmation) OR
2. Patients living in the catchment area of the hospital with invasive salmonellosis confirmed through blood-culture surveillance embedded in routine patient cares

Exclusion Criteria:

* Individuals who do not provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The health care structure in the Democratic Republic of Congo is divided into Health Zones, each subdivided into Health Areas. Each Health Area contains first-line Health Posts and second-line Health Centers, which refer patients requiring advanced care to the Health Zone referral hospital. The study population includes both urban and rural areas and includes approximately 200,000 residents. The greatest distance from remote areas to the tertiary hospital is 80km.
Sampling Method: Probability Sample
Enrollment: 48000 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Typhoid fever | Three years from the time of vaccination
  Blood culture confirmed infection with Salmonella typhi

CONTACTS AND LOCATIONS:
Locations (9):
- Democratic Republic of the Congo (9):
  - Cederi Madimba HC, Kisantu, Bas-Congo Province
  - Gare HC, Kisantu, Bas-Congo Province
  - Kavwaya HC, Kisantu, Bas-Congo Province
  - Kikonka 1 HC, Kisantu, Bas-Congo Province
  - Kintanu Etat HC, Kisantu, Bas-Congo Province
  - Nkandu 1 HC, Kisantu, Bas-Congo Province
  - Nkandu 3 HC, Kisantu, Bas-Congo Province
  - Saint Luc Hospital, Kisantu, Bas-Congo Province
  - Wete HC, Kisantu, Bas-Congo Province